CLINICAL TRIAL: NCT05353348
Title: Effectiveness of Iron Sucrose Combined With rHuEPO and Ascorbic Acid in Improving Perioperative Anaemia in Patients Undergoing Major Cardiac Surgery
Brief Title: Effect of the Combined Programme on Perioperative Anaemia（CPPA）
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0156
Record Dates: First submitted 2022-04-19; First posted 2022-04-29 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Patient Blood Management; Cardiac Surgery; Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferric Oxide, Saccharated; Ascorbic Acid

STUDY DESIGN:
Masking Description: Double blinding is not feasible
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron treatment intervention arm (Experimental): The combination therapy group will receive three treatments consisting of 200 mg/100 ml of iron sucrose IV infusion, 150 IU/Kg of erythropoietin subcutaneously and 2 mg/100 ml of vitamin C IV infusion in the week prior to surgery
  Interventions: Drug: Iron Sucrose, recombinant human erythropoietin, ascorbic acid
- conventional treatment arm (Active Comparator): Treatment in accordance with measures routinely used by the surgeon's team to treat anemia including but not limited to (clinical observation, oral iron supplementation, intravenous iron supplementation, blood transfusion, or other measures) will be documented faithfully by the study team
  Interventions: Procedure: conventional treatment

INTERVENTIONS:
Drug: Iron Sucrose, recombinant human erythropoietin, ascorbic acid — During the 1 week period following admission, 3 consecutive dosing regimens were administered, 200 mg of iron sucrose by intravenous infusion at 8am daily in combination with 150 IU/kg of recombinant human erythropoietin by subcutaneous injection and 2 g of ascorbic acid by intravenous infusion.
  Arms: Iron treatment intervention arm
Procedure: conventional treatment — Treatment in accordance with measures routinely used by the surgeon's team to treat anemia including but not limited to (clinical observation, oral iron supplementation, intravenous iron supplementation, blood transfusion, or other measures) will be documented faithfully by the study team
  Arms: conventional treatment arm

SUMMARY:
We used the preoperative intervention of iron sucrose in combination with human erythropoietin and vitamin C as an innovative combination therapy. This combined treatment strategy aims to improve perioperative anaemia in patients by promoting erythropoiesis and improving iron metabolism. Compared with previous perioperative intravenous iron supplementation, this innovative combination therapy strategy takes into account multiple aspects of iron metabolism as well as the biological mechanisms of erythropoiesis, providing a more comprehensive intervention. Management of perioperative anaemia in previous studies has largely relied on single intravenous iron supplementation therapy, and although this approach has been effective in raising iron levels, its effectiveness may be limited in patients who have impaired iron utilisation or in situations where concurrent stimulation of erythropoiesis is required. The use of iron sucrose in combination with human erythropoietin and vitamin C, on the other hand, is based on an integrative therapeutic concept aimed at providing a more comprehensive response to perioperative anaemia by simultaneously promoting effective iron utilisation and erythropoiesis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Ferritin <300µg/L, transferrin saturation <25%, male 90<Hb<130g/L or female 90<Hb<120g/L
* Elective major cardiac surgery (valve replacement, CABG coronary artery bypass surgery or a combination of both)
* ASA: Grade 1-3
* Signed informed consent

Exclusion Criteria:

1. Allergy or contraindication to iron sucrose or recombinant human erythropoietin or ascorbic acid
2. Patients with a preoperative temperature >37.5 °C or on non-prophylactic antibiotics
3. Pregnancy or breastfeeding stage
4. weight ≤ 50 kg
5. Presence of chronic renal insufficiency, urinary stones, oxalate deposits, gout
6. Chronic liver disease and/or screening alanine transferase/aspartate transferase above normal 3 times or more above the upper limit of the normal range
7. Family history of haemochromatosis, thalassaemia or transferrin saturation > 50%
8. Known history of iron overload
9. Other known causes of anaemia (folic acid or vitamin B12 deficiency or haemoglobinopathies, etc.)
10. Emergency surgery
11. Use of iron, blood transfusion or related anaemia treatment within 12 weeks prior to surgery

Withdrawal criteria:

1. massive blood transfusion (≥ 10 red blood cells (RBC)/24h)
2. Preoperative interventions not performed according to standard
3. Cancellation of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Haemoglobin level on postoperative day 5 | Haemoglobin level on postoperative day 5
  Haemoglobin level on postoperative day 5

SECONDARY OUTCOMES:
Amount of allogeneic blood products used in the perioperative period | From the start of surgery until hospital discharge or postoperative day 30, whichever comes first
  (red blood cells, plasma, platelets)
Effect of combination therapy on changes in perioperative haemoglobin levels | From the start of surgery until hospital discharge or postoperative day 30, whichever comes first
  Pre-intervention versus post-operative haemoglobin
Effect of combination therapy on changes in perioperative ferritin levels | From the start of surgery until hospital discharge or postoperative day 30, whichever comes first
  Pre-intervention versus post-operative ferritin
Effect of combination therapy on changes in perioperative reticulocyte levels | From the start of surgery until hospital discharge or postoperative day 30, whichever comes first
  Magnitude of reticulocyte elevation
Incidence of perioperative acute renal insufficiency | From the start of surgery until hospital discharge or postoperative day 30, whichever comes first
  Postoperative creatinine more than 2 times higher than preoperative or oliguria (<0.5ml/kg/h) within 12 hours
Post-operative intensive care unit stay | From the start of surgery until hospital discharge or postoperative day 30, whichever comes first
  Length of stay in ICU after surgery
Infusion reactions and allergies | From the start of surgery until hospital discharge or postoperative day 30, whichever comes first
  Perioperative allergic events
Incidence of serious adverse events (SAEs) in the perioperative period up to 6 months after surgery | Through study completion, an average of 1.5 year
  Myocardial infarction、Ischemic cerebral infarction、arrhythmia、Deep vein thrombosis of the lower extremity、Pulmonary embolism, etc
All-cause mortality within 6 months of surgery | Through study completion, an average of 1.5 year
  Incidence of mortality
Total length of hospital stay | Through study completion, an average of 1 year
  Total length of hospital stay
Incidence of perioperative infections | Through study completion, an average of 1 year
  Non-prophylactic use of antibiotics
Health Care Costs | From admission until hospital discharge or postoperative day 30, whichever comes first
  All medical costs during hospitalisation
Post-operative hospital readmission rate | Through study completion, an average of 1 year
  Post-operative hospital readmission rate

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- The Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided